CLINICAL TRIAL: NCT02438241
Title: Transcutaneous Electrical Nerve Stimulation Post-thoracic Surgery in a Intensive Care Unit: Randomized Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation Post-thoracic Surgery in a Intensive Care Unit
Acronym: TENS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Hermann Heinrich Husch, Physiotherapist intensive care unit, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36851514.6.0000.5335
Record Dates: First submitted 2015-05-03; First posted 2015-05-08 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-12

CONDITIONS: Thoracic Surgery
Keywords: Pain Measurement; Electric Stimulation; Spirometry; Manometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional physiotherapy Group (Active Comparator): Patients randomized to this group will receive only conventional physiotherapy. The treatment protocol will consist of weathered active exercises to manually lower limbs in bed (triple flexion, abduction and adduction, plantar / dorsiflexion), free active exercises of the upper limbs in the bed (shoulder flexion, shoulder flexion and horizontal functional diagonal shoulder), bronchial hygiene techniques, flow redirection, positive expiratory pressure and ventilatory blowing patterns.
  Interventions: Procedure: Conventional physiotherapy Group
- Placebo TENS Group (Placebo Comparator): Will be held the same procedure as TENS group, except that TENS will be offered to the patient only for 45 seconds, and in the first 30 seconds is reached the sensory threshold of the patient and in the last 15 seconds will turn off the electrical current by 29 remaining period minutes and 15 seconds off.
  Interventions: Procedure: Placebo TENS group
- TENS group (Experimental): Patients randomized to this group will receive conventional physical therapy for the control group, and the end of that service, will be applied TENS. TENS is accomplished through the use of an electrical stimulation device with symmetrical biphasic current pulse. The following parameters are used: frequency: 100 Hz, pulse width: 100 µs, intensity to the greatest sensory threshold of the patient and total session time: 30 minutes. Self-adhesive electrodes will be used (Valutrode, size 5x9 cm) to be positioned in the posterolateral portion of the chest to 2 cm skin incision both upper and lower.
  Interventions: Procedure: TENS Group

INTERVENTIONS:
Procedure: Conventional physiotherapy Group — Patients randomized to this group will receive only conventional physiotherapy. The treatment protocol Control Group, will consist of weathered active exercises to manually lower limbs in bed (triple flexion, abduction and adduction, plantar / dorsiflexion), free active exercises of the upper limbs in the bed (shoulder flexion, shoulder flexion and horizontal functional diagonal shoulder), bronchial hygiene techniques, flow redirection, positive expiratory pressure and ventilatory blowing patterns.
  Arms: Conventional physiotherapy Group
Procedure: TENS Group — Patients randomized to this group will receive conventional physical therapy (the treatment protocol Control Group), and the end of that service, will be applied TENS. TENS is accomplished through the use of an electrical stimulation device with symmetrical biphasic current pulse. The following parameters are used: frequency: 100 Hz, pulse width: 100 µs, intensity to the greatest sensory threshold of the patient and total session time: 30 minutes. Self-adhesive electrodes will be used (Valutrode, size 5x9 cm) to be positioned in the posterolateral portion of the chest to 2 cm skin incision both upper and lower.
  Arms: TENS group
Procedure: Placebo TENS group — Patients randomized to this group will receive conventional physical therapy (the treatment protocol Control Group), will be held the same procedure as TENS group, except that TENS will be offered to the patient only for 45 seconds, and in the first 30 seconds is reached the sensory threshold of the patient and in the last 15 seconds will turn off the electrical current by 29 remaining period minutes and 15 seconds off.
  Arms: Placebo TENS Group

SUMMARY:
Introduction: Pain is an important factor of increase of morbidity and mortality in patients undergoing surgical procedures include thoracotomy. There are different methods of analgesia in postoperative thoracic surgery, ranging from systemic analgesia with opioids, as well as local anesthetics block (intrapleural, extrapleural, intercostal cryoanalgesia, etc.) in addition to spinal blocks and Epidural blocks. In the pharmacological analgesia, electroanalgesia has been proposed as an adjunctive treatment for the relief of postoperative pain. Rationale: noting the lack of data in the literature regarding the use of this physical therapy technique in order to reduce the pain in the postoperative period of thoracic surgery and its consequences, it is relevant to the realization of a new randomized controlled trial (RCT) to evaluate the effects of transcutaneous electrical nerve (TENS) in the post - thoracic surgery on pain, pulmonary function and strength respiratory muscle. Objective: To evaluate the effects of TENS on pain, respiratory muscle strength and lung function in postoperative thoracic surgery in a Intensive Care Unit. Method: The subjects included will be randomized into three groups randomly: control group (CG) that will hold only conventional physical therapy, TENS group (EG) that will hold the application of TENS associated with conventional physical therapy, TENS placebo group (GP) who will perform the application of TENS placebo to conventional therapy. All groups carry out the assessments (digital manometer, spirometry, visual analog pain scale) in the preoperative period, postoperative Immediate / pre-intervention and at the end of treatment (discharge from the intensive care unit), except for the pain that will be evaluated before and after each intervention session. All patients receive physical therapy three times a day (morning, afternoon and evening) during hospitalization in the intensive care unit. Intervention: The conventional group will receive conventional therapy for hospital service. The TENS group will receive conventional therapy and the end of that service, will be applied TENS for 30 minutes. The placebo TENS group will receive the conventional physical therapy and the end of the service will be installed TENS placebo, during this period the patient receives electrical stimulation for 45 seconds, shutting down at the end of this time and held position as TENS group.

DETAILED DESCRIPTION:
An evaluation of the patient will be held in the preoperative through a standardized form containing all personal data and information regarding the history and physical examination. At this time, the patient, after reading and removal of doubts, or his guardian sign the Informed Consent making clear consent to participate. After the arrival of the surgical patient will evaluate eligibility criteria. Subjects included will be randomized into three groups randomly: control group (CG) that will hold only conventional physical therapy, TENS group (EG) that will hold the application of TENS associated with conventional physical therapy, TENS placebo group (GP) that will hold the application TENS placebo to conventional therapy. All groups carry out the assessments described below in the preoperative period, in the immediate post-operative / pre-intervention (up to 6 hours after arrival in the intensive care unit) and the end of treatment (discharge from the intensive care unit), except for the pain that will be evaluated before and after each intervention session. All patients receive physical therapy three times a day (morning, afternoon and evening) during their stay in the intensive care unit. Pain assessment: To measure the painful sensation, visual analogue scale pain will be used. Evaluation of lung function: Pulmonary function is assessed by spirometry with a portable digital spirometer Sibelmed brand, Datospir micro c model, with the objective of obtaining the lung volume and capacity. The patient is positioned in the bed (head elevated at 90º, extended legs, nasal clips in the patient (ensures optimal sealing), is positioned in the mouth patient requested a maximal inspiration followed by a maximum and sustained expiration through the mouth. During exhalation the patient will be encouraged verbally to achieve your best performance. As recommended by the American Thoracic Society and European Respiratory Society and based on the reproducibility and eligibility criteria, three maneuvers will be performed (variability of 0.150L) and considered the best curve for study. They will be obtained the forced vital capacity values (FVC), forced expiratory volume in one second (FEV1), FEV1 / FVC, peak expiratory flow and forced expiratory flow between 25 and 75% of FVC curve. The values will be recorded in absolute units of measurement and percentage of predicted. Due to the high variability between operators, this evaluation will be performed by the same researcher. Evaluation of respiratory muscle strength: To evaluate the inspiratory and expiratory muscle strength will be used, respectively, measurements of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) through a digital manometer Globalmed make, model MVD300. The patient is positioned in the bed (headboard raised to 90 °), extended legs and a nose clip. The test is repeated 6 times with one-minute interval between each attempt, is considered the highest value since there is no difference greater than 10% between the two highest values. The MIP will be determined, based on the residual volume, the deep breath against the occluded circuit and the MEP will be obtained, starting from the total lung capacity, the expiration forced against the machine's nozzle. For analysis of the results will be considered absolute and in percentage of predicted by the equations proposed by Neder et al. Assessing the amount of medication administered: Patients from surgery can come with two types of fixed analgesia: epidural catheter or paravertebral catheter. These catheters can come up with: bupivacaine fentanyl; ropivacaine fentanyl. In addition the catheters are prescribed acetaminophen, dipyrone, tramadol, morphine. The type of fixing is controlled analgesia, dosage and dosage for each investigator assessment, furthermore all be checked to check prescriptions adjunct administered throughout the day.

Interventions TENS group: Patients randomized to this group will receive conventional physical therapy for the control group, and the end of that service, will be applied TENS. TENS is accomplished through the use of an electrical stimulation device with symmetrical biphasic current pulse. The following parameters are used: frequency: 100 Hz, pulse width: 100 µs, intensity to the greatest sensory threshold of the patient and total session time: 30 minutes. Self-adhesive electrodes will be used (Valutrode, size 5x9 cm) to be positioned in the posterolateral portion of the chest to 2 cm skin incision both upper and lower.

Placebo TENS group: Will be held the same procedure as TENS group, except that TENS will be offered to the patient only for 45 seconds, and in the first 30 seconds is reached the sensory threshold of the patient and in the last 15 seconds will turn off the electrical current by 29 remaining period minutes and 15 seconds off.

Control group: Patients randomized to this group will receive only conventional physiotherapy. The treatment protocol will consist of weathered active exercises to manually lower limbs in bed (triple flexion, abduction and adduction, plantar / dorsiflexion), free active exercises of the upper limbs in the bed (shoulder flexion, shoulder flexion and horizontal functional diagonal shoulder), bronchial hygiene techniques, flow redirection, positive expiratory pressure and ventilatory blowing patterns.

ELIGIBILITY:
Inclusion Criteria:

* Will be included patients between 30 and 75 years;
* Both sexes;
* Post-thoracic surgery with posterolateral thoracotomy incision for pulmonary resection (Bullectomy, segmentectomy, lobectomy, pneumonectomy);
* Evaluated between 4-6 hours after entry into the intensive care unit;
* Hemodynamic stability (mean arterial pressure between 60 mmHg and 100 mmHg, heart rate between 50 bpm and 110 bpm, peripheral saturation greater than 90%);
* Patients who have liquid drainage chest tubes in less than 300 ml for six hours;
* Scale agitation-sedation Richmond (RASS) between -1 and +1;
* Prescription physical therapy;
* Have epidural or Paravertebral catheter;
* Agree to participate in the study by signing the Informed Consent and Informed (IC ).

Exclusion Criteria:

* Not intubated with up to 6 hours in the immediate postoperative period;
* Primary pulmonary disease not rise (cardiovascular, neurological diseases);
* Hemodynamic instability (with pressure mean blood less than 60 mmHg or greater 100 mmHg, heart rate less than 49 bpm and greater than 111 bpm, reduced peripheral saturation of 90%);
* Patients who have the upper drainage liquid drains to 300 ml for six hours;
* Scale agitation-sedation Richmond (RASS) between -5 and -2, and agitated / aggressive patients, scale agitation-sedation Richmond RASS +2 and +4;
* Prescribing physical therapy;
* Without epidural or paravertebral catheter;
* Patients who do not accept the study, not collaborative and do not sign the informed consent form.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Assess the pain of change in postoperative thoracic surgery | 3 days
  It will be used a visual analogous scale to assess pain after each service physiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, doctor, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Irmandade Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Landreneau RJ, Pigula F, Luketich JD, Keenan RJ, Bartley S, Fetterman LS, Bowers CM, Weyant RJ, Ferson PF. Acute and chronic morbidity differences between muscle-sparing and standard lateral thoracotomies. J Thorac Cardiovasc Surg. 1996 Nov;112(5):1346-50; discussion 1350-1. doi: 10.1016/S0022-5223(96)70150-2. PMID 8911333
- [Result] Savage C, McQuitty C, Wang D, Zwischenberger JB. Postthoracotomy pain management. Chest Surg Clin N Am. 2002 May;12(2):251-63. doi: 10.1016/s1052-3359(02)00011-x. PMID 12122825
- [Result] Kavanagh BP, Katz J, Sandler AN. Pain control after thoracic surgery. A review of current techniques. Anesthesiology. 1994 Sep;81(3):737-59. doi: 10.1097/00000542-199409000-00028. No abstract available. PMID 8092520
- [Result] Boisseau N, Rabary O, Padovani B, Staccini P, Mouroux J, Grimaud D, Raucoules-Aime M. Improvement of 'dynamic analgesia' does not decrease atelectasis after thoracotomy. Br J Anaesth. 2001 Oct;87(4):564-9. doi: 10.1093/bja/87.4.564. PMID 11878725
- [Result] Benedetti F, Amanzio M, Casadio C, Cavallo A, Cianci R, Giobbe R, Mancuso M, Ruffini E, Maggi G. Control of postoperative pain by transcutaneous electrical nerve stimulation after thoracic operations. Ann Thorac Surg. 1997 Mar;63(3):773-6. doi: 10.1016/s0003-4975(96)01249-0. PMID 9066400
- [Result] Yegin A, Erdogan A, Kayacan N, Karsli B. Early postoperative pain management after thoracic surgery; pre- and postoperative versus postoperative epidural analgesia: a randomised study. Eur J Cardiothorac Surg. 2003 Sep;24(3):420-4. doi: 10.1016/s1010-7940(03)00345-2. PMID 12965314
- [Result] Grant RP. Con: every postthoracotomy patient does not deserve thoracic epidural analgesia. J Cardiothorac Vasc Anesth. 1999 Jun;13(3):355-7. doi: 10.1016/s1053-0770(99)90277-x. No abstract available. PMID 10392691
- [Result] Baidya DK, Khanna P, Maitra S. Analgesic efficacy and safety of thoracic paravertebral and epidural analgesia for thoracic surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2014 May;18(5):626-35. doi: 10.1093/icvts/ivt551. Epub 2014 Jan 31. PMID 24488821
- [Result] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Result] Chandra A, Banavaliker JN, Das PK, Hasti S. Use of transcutaneous electrical nerve stimulation as an adjunctive to epidural analgesia in the management of acute thoracotomy pain. Indian J Anaesth. 2010 Mar;54(2):116-20. doi: 10.4103/0019-5049.63648. PMID 20661348
- [Result] Erdogan M, Erdogan A, Erbil N, Karakaya HK, Demircan A. Prospective, Randomized, Placebo-controlled Study of the Effect of TENS on postthoracotomy pain and pulmonary function. World J Surg. 2005 Dec;29(12):1563-70. doi: 10.1007/s00268-005-7934-6. PMID 16331341
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Derived] Husch HH, Watte G, Zanon M, Pacini GS, Birriel D, Carvalho PL, Kessler A, Sbruzzi G. Effects of Transcutaneous Electrical Nerve Stimulation on Pain, Pulmonary Function, and Respiratory Muscle Strength After Posterolateral Thoracotomy: A Randomized Controlled Trial. Lung. 2020 Apr;198(2):345-353. doi: 10.1007/s00408-020-00335-4. Epub 2020 Feb 8. PMID 32036406
- See also: Estimulação elétrica nervosa transcutânea no pós-operatório de cirurgia torácica: revisão sistemática e metanálise de estudos randomizados — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0102-76382012000100012